CLINICAL TRIAL: NCT03911245
Title: Our Experience About Limb and Pelvic Osteosarcoma in Patients Older Than 40 Years and Comparative Study With the Age Group < 40 Years. Prognostic Factors, Survival, Amputation Rate and Limb Salvage Surgery After Neoadjuvant Chemotherapy
Brief Title: Osteosarcoma in Patients Older Than 40 Years. Prognostic Factors and Survival
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-OST-2017-67
Record Dates: First submitted 2019-03-03; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Medical Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with age equal or older than 40 years
  Interventions: Other: Retrospective study. Analyze of data in medical records
- Patients with age less than 40 years
  Interventions: Other: Retrospective study. Analyze of data in medical records

INTERVENTIONS:
Other: Retrospective study. Analyze of data in medical records — Retrospective study. Analyze of data in medical records

SUMMARY:
The purpose of this work is to carry out an exhaustive analysis of the characteristics of osteosarcoma in patients with an age equal to or greater than 40 years, in the Hospital de la Santa Creu and Sant Pau in Barcelona, during the years 1986-2016, with the objective to establish the factors that determine the disease and survival, as well as to evaluate the rates of limb salvage and amputation after neodyuvant chemotherapy. With the result of the results, the report of osteosarcoma and the age less than 40 years, with the aim of providing new information that is related to the appearance of osteosarcoma is available from 40 years.

DETAILED DESCRIPTION:
The main objectives of this study are the following:

* Describe the prognostic factors of osteosarcoma in patients aged 40 years or older, treated at the Hospital de la Santa Creu and Sant Pau in Barcelona during the years 1986-2016, as well as overall survival and disease-free survival.
* Quantify the frequency of limb salvage surgery and amputation, determining the influence of the use of neoadjuvant chemotherapy in the definitive therapeutic management.
* Compare the results obtained with a group formed patients with a range of less than 40 years, diagnosed and treated with osteosarcoma at the Hospital de la Santa Creu i Sant Pau in Barcelona during the same period of years.

The secondary objectives of this study are the following:

* Analyze the frequency of occurrence of local recurrence.
* Determine postoperative complications.
* Evaluate the frequency of distant spread of the disease.
* Describe the characteristics of the group of patients in the study.
* Demonstrate that the incidence of osteosarcoma in adulthood is increasing over the years.
* Determine predisposing factors or lesions to the appearance of osteosarcoma not described in the literature.

ELIGIBILITY:
First age group (equal or> 40 years old):

* Inclusion criteria:

  * Osteosarcoma localized in axial skeleton or limbs, diagnosis confirmed by performing a biopsy of the lesion in the Hospital of Santa Creu i Sant Pau, and subsequent histological analysis by the Pathological Anatomy Service of the same center, or, by histological review of the sample from the biopsy performed in the reference center of patients from other hospitals.
  * Age equal to or greater than 40 years.
  * Minimum follow-up of 12 months. The patients included in the study have met all the inclusion criteria.
* Exclusion criteria:

  * Osteosarcomas from other locations (head, neck, thorax and cervical, dorsal or lumbosacral spine).
  * Age less than 40 years.
  * Follow-up less than 12 months.
  * Patients who present as a single surgical intervention, and therefore, osteosarcoma was not treated surgically in a definitive manner.
  * Patients in whom there is an inconsistency between the histological diagnosis of the biopsy and the resection piece, that is, the diagnosis after the definitive study of the resection piece has not corresponded to the osteosarcoma, although it is outside the histological study of the bone biopsy.
  * Patients who have undergone a surgical treatment of their tumor lesion, except in the diagnostic biopsy, in another hospital center.

Second age group (<40 years):

• Inclusion criteria:

* Osteosarcoma localized in axial skeleton or limbs, diagnosis confirmed by performing a biopsy of the lesion in the Hospital of Santa Creu i Sant Pau, and subsequent histological analysis by the Pathological Anatomy Service of the same center, or, by histological review of the sample obtained from the biopsy performed in the reference center of patients from other hospitals.
* Age less than 40 years for the first age group.
* Minimum follow-up of 12 months.

The patients included in the study have met all the inclusion criteria.

• Exclusion criteria:

* Osteosarcomas from other locations (head, neck, thorax and cervical, dorsal or lumbosacral spine).
* Age equal to or greater than 40 years.
* Follow-up less than 12 months.
* Patients subjected to a biopsy as the only surgical intervention, and that therefore, osteosarcoma was not definitively treated surgically.
* Patients in whom there is an incongruence between the histological diagnosis of the biopsy and the resection piece, that is, the diagnosis after the definitive study of the resection piece has not corresponded to that of osteosarcoma, although initially it was after the study Histological examination of the bone biopsy.
* Patients who have undergone a surgical treatment of their tumor lesion, except for the diagnostic biopsy, in another hospital center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with osteosarcoma located in the extremities or pelvis.
  Number of subjects over 40 years: 37 patients. Number of subjects under 40 years old: 100 patients.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Prognostic factors of osteosarcoma | 1 year
  The impact of prognostic factors was assessed using the log-rank test in univariate analysis. Multivariate analysis was undertaken using the Cox proportional hazards method, with variables chosen using logistic regression with a backward stepwise approach. Relative risks were calculated using the Cox proportional hazards model with only the noted covariate in the model. A p value <0.05 was considered significant. Confidence intervals of 95 % were calculated for statistical parameters. Statistical analysis was performed using SPSS 24.0 for Windows.
Survival of osteosarcoma | 1 year
  Overall survival (OS) was defined as the period from date of diagnosis to date of death or last follow-up, and was calculated using Kaplan-Meier survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Almenara, Principal Investigator — Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bacci G, Longhi A, Versari M, Mercuri M, Briccoli A, Picci P. Prognostic factors for osteosarcoma of the extremity treated with neoadjuvant chemotherapy: 15-year experience in 789 patients treated at a single institution. Cancer. 2006 Mar 1;106(5):1154-61. doi: 10.1002/cncr.21724. PMID 16421923
- [Result] Joo MW, Shin SH, Kang YK, Kawai A, Kim HS, Asavamongkolkul A, Jeon DG, Kim JD, Niu X, Tsuchiya H, Puri A, Wang EH, Chung SH, Chung YG. Osteosarcoma in Asian Populations Over the Age of 40 Years: A Multicenter Study. Ann Surg Oncol. 2015 Oct;22(11):3557-64. doi: 10.1245/s10434-015-4414-6. Epub 2015 Feb 13. PMID 25676843
- [Result] Longhi A, Errani C, Gonzales-Arabio D, Ferrari C, Mercuri M. Osteosarcoma in patients older than 65 years. J Clin Oncol. 2008 Nov 20;26(33):5368-73. doi: 10.1200/JCO.2007.14.9104. Epub 2008 Sep 22. PMID 18809616
- [Result] Iwata S, Ishii T, Kawai A, Hiruma T, Yonemoto T, Kamoda H, Asano N, Takeyama M. Prognostic factors in elderly osteosarcoma patients: a multi-institutional retrospective study of 86 cases. Ann Surg Oncol. 2014 Jan;21(1):263-8. doi: 10.1245/s10434-013-3210-4. Epub 2013 Aug 23. PMID 23975321
- [Result] Grimer RJ, Cannon SR, Taminiau AM, Bielack S, Kempf-Bielack B, Windhager R, Dominkus M, Saeter G, Bauer H, Meller I, Szendroi M, Folleras G, San-Julian M, van der Eijken J. Osteosarcoma over the age of forty. Eur J Cancer. 2003 Jan;39(2):157-63. doi: 10.1016/s0959-8049(02)00478-1. PMID 12509946
- [Result] Carsi B, Rock MG. Primary osteosarcoma in adults older than 40 years. Clin Orthop Relat Res. 2002 Apr;(397):53-61. doi: 10.1097/00003086-200204000-00008. PMID 11953595